CLINICAL TRIAL: NCT05472168
Title: SNEEX - Impact of Olfactory Odour StimulatioN on Energy EXpenditure
Brief Title: Impact of Olfactory Odour StimulatioN on Energy EXpenditure
Acronym: SNEEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Katharina Timper, Principal Investigator, Prof. Dr. med., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Timper_Olfactory_2022
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese (Other): Age 18-55 years Obesity (BMI ≥30 kg/m2) Written informed consent Normosmia (defined by sniffing Sticks test)
  Interventions: Other: Olfactory Stimulation
- Lean (Other): Age 18-55 years Lean (BMI 18-25 kg/m2) Written informed consent Normosmia (defined by sniffing Sticks test)
  Interventions: Other: Olfactory Stimulation

INTERVENTIONS:
Other: Olfactory Stimulation — Participants are exposed to different odours and energy expenditure is assessed via indirect calorimetry.
  Other Names: Different odours

SUMMARY:
In this preliminary short-term study it is investigated, whether a short olfactory stimulation with distinct odours impacts energy expenditure in patients with obesity and lean patients.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-55 years

  * Obesity (BMI ≥30 kg/m2) and Lean (BMI 18-25 kg/m2)
  * Written informed consent
  * Normosmia (defined by sniffing Sticks test)

Exclusion Criteria:

* • Chronic or acute sinusitis

  * Surgical intervention of the nasal cavity or the paranasal sinus
  * Known allergy to odors used in the study
  * Smokers
  * Current illicit drug abuse including daily marijuana and cannabidiol (CBD) consumption (alcohol ≤2 drinks per day allowed)
  * Any kind of severe chronic disease (e.g. severe heart failure, active cancer disease)
  * Diabetes mellitus
  * Treatment with insulin sensitizing drugs including Glucagon-like Peptide (GLP)-1 analogues within the last 3 months
  * History of neurodegenerative diseases, severe head trauma
  * Severe renal impairment (e.g. estimated glomerular filtration rate <30 ml/min/m2)
  * Known liver cirrhosis or other severe liver impairment
  * Use of any kind of decongestant more than twice a week
  * Use of cortisone-containing nasal spray within the last 3 months
  * Acute upper respiratory tract infection
  * Uncontrolled dysthyroidism
  * Uncontrolled hypertension
  * Regular use of psychopharmaceutic drugs
  * Study participants aims to start a new diet or exercise program during the study
  * Bariatric surgery
  * Pregnancy/Lactation
  * Onset of climacteric symptoms within one year (e.g. hot flashes and/or diaphoresis) OR initiation of hormonal replacement therapy in the last three months
  * Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
  * Participation in an interventional study within the last 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Energy Expenditure | 6 hours
  change in energy expenditure as assessed via calorimetry after olfactory stimulation with different odours.

SECONDARY OUTCOMES:
Energy Expenditure, Additional Odours | 6 hours
  Change in energy expenditure as assessed via calorimetry after olfactory stimulation with Different odours
Heart Rate | 6 hours
  change in heart rate variability upon olfactory stimulation with different odors as assessed via continuous ECG
Blood Pressure | 6 hours
  Change in blood pressure upon olfactory stimulation with different odors as assessed via a blood pressure cuff at the upper arm according to Riva Rocci
Metabolic Parameters | 6 hours
  Change in metabolic blood parameters upon acute olfactory stimulation with different odours
Glucose Levels | 6 hours
  change in interstitial fluid glucose levels upon olfactory stimulation with different odours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland